CLINICAL TRIAL: NCT04059289
Title: Intermediate Vision in a Driving Simulator Environment: Comparison of the New J&J EYHANCE IOL With a Conventional Monofocal IOL
Brief Title: Intermediate Vision in a Driving Simulator Environment: Comparison of the J&J EYHANCE With a Conventional Monofoc. IOL
Acronym: JJ-EYHANCE
Status: Completed | Type: Observational
Sponsor: Aalen University (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: JJ-EY-AA_1
Record Dates: First submitted 2019-08-08; First posted 2019-08-16 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2019-08

CONDITIONS: Lenses, Intraocular; Pseudophakia; Near Vision; Driving
Keywords: glare; contrast sensitivity; driving simulator; intermediate visual acuity; pseudophakia; posterior chamber intraocular lenses; benchmark; straylight; nighttime driving
MeSH Terms: conditions — Pseudophakia; Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Two types of intraocular lenses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intraocular lens type I: Tecnis EYHANCE IOL (Johnson & Johnson, New Brunswick/USA)
  Interventions: Other: Posterior chamber intraocular lens (IOL)
- Intraocular lens type II: Clareon IOL (Alcon Pharma. Freiburg/FRG)
  Interventions: Other: Posterior chamber intraocular lens (IOL)

INTERVENTIONS:
Other: Posterior chamber intraocular lens (IOL) — This is NOT an interventional study; the intervention (surgical procedure) has been performed PRIOR to the inclusion in this study
  Other Names: Tecnis EYHANCE IOL (Johnson & Johnson, New Brunswick/USA); Clareon IOL (Alcon Pharma. Freiburg/FRG)

SUMMARY:
To compare (low contrast) visual acuity (VA) and contrast sensitivity (CS) - both at intermediate distances under nighttime driving conditions in a driving simulator between patients with bilateral EYHANCE IOLs OR bilateral conventional monofocal IOLs. Visual function testing in the driving simulator will be assessed without AND with (static) glare.

Additionally: Assessment of individual response times, scanpath characteristics, evaluation of test retest reliability and self-evaluation of (intermediate) vision and visual impairment related to glare.

DETAILED DESCRIPTION:
To compare (low contrast) visual acuity (VA) and contrast sensitivity (CS) - both at intermediate distances under nighttime driving conditions in a driving simulator between patients with bilateral EYHANCE IOLs OR bilateral conventional monofocal IOLs. Visual function testing in the driving simulator will be assessed without AND with (static) glare.

Additionally: Assessment of individual response times, scanpath characteristics, evaluation of test retest reliability and self-evaluation of (intermediate) vision and visual impairment related to glare.

Simulator

Patients are instructed to drive with a constant speed of 40 km/h on a virtual parcours (straight lane). For testing of either (low contrast) visual acuity or contrast sensitivity, 8-position LANDOLT C's are presented at three locations (within the simulator car, AUDI A4, Ingolstadt/FRG):

(i) At the center of the instrument panel (distance 0.xx m) (ii) At the center of the navigation monitor (y.yy m) (iii) At the center of the rear monitor (z.zz m) A high resolution acoustic attention guidance for immediate gaze direction of the patients towards the three above-mentioned visual stimulus locations (i-iii) is mandatory.

Patients responses are recorded and response times can be extracted from the recordings.

Clinical ophthalmological-optical examinations

* Medical/ophthalmological history
* (Uncorrected and Best-corrected) visual acuity (RE,LE,BE) with remote and intermediate (66cm) 8 position LANDOLT C's.
* LANG I stereotest (near distance)
* Ocular alignment & ocular motility
* Efferent & afferent pupillomotor status
* Mesopic contrast sensitivity without/with glare (Optovist, VISTEC Inc./Olching/FRG)
* Intraocular straylight perception (Q-Quant, OCULUS Inc, Wetzlar/FRG)
* Slit lamp (anterior segment)
* Ophthalmoscope (central fundus and fixation)

  * Primary objectives: log visual acuity (logVA) at preset low contrast level of 1:2.7 (logCS = 0.2) AND log contrast sensitivity (logCS) at a preset visual acuity level of 0.1 = 2/20)
  * Secondary objectives: test retest reliability (as operationalized by LOA = limits of agreement) AND response time (i.e. time interval between onset of stimulus presentation and final response) AND scanpath characteristics (fixation duration, fixation stability, annotation to regions of interest; saccade amplitude) self-evaluation (questionnaire, using visual analogue scales = VAS)

SHAPIRO WILK test (statistical testing for proving/disproving normal distribution) Descriptive statistics (either MEAN, standard deviation, in case of normally distributed data - else, MEDIAN, inter-quartile range (IQR).

Assessment of test/retest reliability: BLAND ALTMAN plots, limits of agreement (LOA) Between-group comparison: t-test (unpaired samples), in case of normally distributed data - else, WILCOXON signed-rank test

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* S.p. (at least two months post surgery) bilateral uneventful IOL surgery (bilateral implantation of either EYHANCE IOL OR monofocal IOL)
* Ophthalmological history normal, except cataract and uneventful IOL surgery
* Distant visual high-contrast acuity > 20/25 in either eye
* Normal stereopsis (all figures of the LANG I random dot stereo test correctly recognized)

Exclusion Criteria:

* Age below 18 years
* Chronic eye disease (except cataract)
* History of ocular surgery (except complication-free IOL surgery)
* Visual pathway lesions
* Strabismus

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects of male or femal gender above the age of 18 years at least two months post surgery after bilateral uneventful IOL surgery (bilateral implantation of either EYHANCE IOL OR monofocal IOL)
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
logVA | at least two months after uneventful intraocular lens implantation
  logarithm of visual acuity at preset low contrast level of 1:2.7 (logCS = 0.2)
logCS | at least two months after uneventful intraocular lens implantation
  logarithm of contrast sensitivity at a preset visual acuity level of 0.1 (= 2/20)

SECONDARY OUTCOMES:
Reproducibilities of logVA | at least two months after uneventful intraocular lens implantation
  as operationalized by LOA (limits of agreement)
Resonse times of logCS | at least two months after uneventful intraocular lens implantation
  time interval between onset of stimulus presentation amd final response
Scanpath characteristics (I) | at least two months after uneventful intraocular lens implantation
  fixation duration
Scanpath characteristics (II) | at least two months after uneventful intraocular lens implantation
  fixation stability
Scanpath characteristics (III) | at least two months after uneventful intraocular lens implantation
  annotation to regions of interest (ROIs)
Scanpath characteristics (IV) | at least two months after uneventful intraocular lens implantation
  saccade amplitude
Self-evaluation (questionnaire) (i) distant vision with best distant correction | at least two months after uneventful intraocular lens implantation
  Distant vision (self-eval., vis. analogue scales: 0 = unsatisfactory ... 10 = optimal)
Self-evaluation (questionnaire) (i) intermediate vision with best distant correction | at least two months after uneventful intraocular lens implantation
  Intermed. vision (self-eval., vis. analog. scales: 0 = unsatisfactory ... 10 = optimal)
Self-evaluation (questionnaire) (i) mesopic vision with best distant correction | at least two months after uneventful intraocular lens implantation
  Mesopic vision (self-eval., vis. analog. scales: 0 = unsatisfactory ... 10 = optimal)
Self-evaluation (questionnaire) (i) glare sensitivity with best distant correction | at least two months after uneventful intraocular lens implantation
  Glare sensitivity (self-eval., vis. analog. scales: 0 = unsatisfactory ... 10 = optimal)
Self-evaluation (questionnaire) (i) General post-op vision with best distant corr. | at least two months after uneventful intraocular lens implantation
  Post-op vision (self-eval., vis. analog. scales: 0 = unsatisfactory ... 10 = optimal)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Applied Sciences, Study Course Ophthalmic Optics, Aalen, Baden-Wurttemberg, Germany